CLINICAL TRIAL: NCT04322019
Title: Prescription Strategies of Amikacin in Intensive Care Patients on Renal Replacement Therapy: an Observational Prospective Multicenter Study
Acronym: AMIDIAL-ICU
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO20032
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Amikacin Treatment
Keywords: Amikacin; intensive care; renal replacement therapy; prescription strategy,; monitoring strategy
MeSH Terms: interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "Amikacin treatment" group: Intensive care patients on renal replacement therapy with Amikacin treatment
  Interventions: Other: Data record

INTERVENTIONS:
Other: Data record — Data record

SUMMARY:
Amikacin is the aminoglycoside of choice for treatment of severe infections in intensive care. An achievement of its objectives in pharmacokinetics and pharmacodynamics is difficult in intensive care patients because of modification of their volume of distribution and renal clearance. Acute renal failure requiring renal replacement therapy is frequent in intensive care. Extrarenal purification modalities (continuous versus intermittent, type of dialysis membrane), which can influence amikacin clearance, are multiple and teams dependent. Guidelines of good practice for Amikacin in intensive care patients do not exist.

DETAILED DESCRIPTION:
The aim of this study is to describe strategies of prescription and monitoring of Amikacin in intensive care patients on renal replacement therapy.

ELIGIBILITY:
inclusion criteria :

* patients in intensive care
* patients on extrarenal replacement
* patients with Amikacin treatment
* patients accepting to participate in the study

exclusion criteria :

* patients less than 18 years old
* pregnant women
* patients with Amikacin treatment in the previous 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients on renal replacement therapy with Amikacin treatment
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Measurement of maximum concentration observed | Day 0
  Monitoring of Amikacin treatment using measurement of maximum concentration observed performed or not

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France